CLINICAL TRIAL: NCT03353753
Title: A Phase 3, INterVentional, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of DCC-2618 In Patients With AdvanCed Gastrointestinal Stromal TUmorS Who Have Received Treatment With Prior Anticancer Therapies
Brief Title: Phase 3 Study of DCC-2618 vs Placebo in Advanced GIST Patients Who Have Been Treated With Prior Anticancer Therapies
Acronym: INVICTUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Deciphera Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DCC-2618-03-001
Record Dates: First submitted 2017-11-20; First posted 2017-11-27 (Actual); Results first posted 2021-04-23 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — ripretinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): 150 mg QD DCC-2618
  Interventions: Drug: DCC-2618
- Arm 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: DCC-2618 — Oral KIT/PDGFRA kinase inhibitor
  Other Names: ripretinib
  Arms: Arm 1
Drug: Placebo Oral Tablet — Placebo
  Arms: Arm 2

SUMMARY:
This is a 2-arm, randomized, placebo-controlled, double-blind, international, multicenter study comparing the efficacy of ripretinib (DCC-2618) to placebo in patients who have received treatment with prior anticancer therapies. Prior anticancer therapies must include imatinib, sunitinib, and regorafenib (3 prior therapies). Approximately 120 patients were randomized in a 2:1 ratio to ripretinib 150 mg QD or placebo

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of GIST
2. Patients must have progressed on imatinib, sunitinib, and regorafenib or have documented intolerance to any of these treatments.
3. ECOG PS of 0 to 2 at screening.
4. Able to provide an archival tumor tissue sample if no anticancer therapy was administered since the sample was collected; otherwise, a fresh tumor tissue sample is required prior to the first dose of study drug.
5. Female patients of childbearing potential must have a negative serum beta-human chorionic gonadotrophin (β-hCG) pregnancy test at screening and negative urine pregnancy test at Cycle 1 Day 1 prior to the first dose of study drug.
6. Patients of reproductive potential must agree to follow the contraception requirements.
7. The patient is capable of understanding and complying with the protocol and has signed the informed consent document. A signed informed consent form must be obtained before any study-specific procedures are performed.
8. At least 1 measurable lesion according to modified RECIST Version 1.1 (non-nodal lesions must be ≥1.0 cm in the long axis or ≥double the slide thickness in the long axis) within 21 days prior to the first dose of study drug.
9. Adequate organ function and bone marrow reserve as indicated by the following laboratory assessments performed at screening.

   * Absolute neutrophil count ≥1000/uL
   * Hemoglobin ≥8 g/dL
   * Platelet count ≥75,000/uL
   * Total bilirubin ≤1.5 x the upper limit of normal (ULN)
   * Aspartate transaminase or alanine transaminase ≤3 x ULN (≤5x ULN in the presence of hepatic metastases)
   * Serum creatinine ≤1.5 x ULN or creatinine clearance ≥50 mL/min based on either urine collection or Cockcroft Gault estimation.
   * Prothrombin time (PT) or international normalized ratio (INR) or partial thromboplastin time ≤1.5 x ULN. Patients on a stable, maintenance regimen of anticoagulant therapy for at least 30 days prior to study drug administration may have PT/INR measurements >1.5 x ULN if, in the opinion of the Investigator, the patient is suitable for the study. An adequate rationale must be provided to the Sponsor prior to randomization.
10. Resolution of all toxicities from prior therapy to ≤Grade 1 (or baseline) within 1 week prior to the first dose of study drug (excluding alopecia and ≤Grade 3 clinically asymptomatic lipase, amylase, and creatine phosphokinase laboratory abnormalities).

Exclusion Criteria:

1. Treatment with anticancer therapy, including investigational therapy, or investigational procedures within 14 days or 5 x the half-life (whichever is longer) prior to the first dose of study drug. For prior biological therapies, eg, monoclonal antibodies with a half-life longer than 3 days, the interval must be at least 28 days prior to the first dose of study drug.
2. Prior treatment with DCC-2618
3. Prior or concurrent malignancy whose natural history or treatment have the potential to interfere with the safety or efficacy assessment of DCC-2618. Patients receiving adjuvant cancer treatment are not eligible if those medications are potentially active against GIST or excluded per protocol.
4. Patient has known active central nervous system metastases.
5. New York Heart Association class II - IV heart disease, active ischemia or any other uncontrolled cardiac condition such as angina pectoris, clinically significant cardiac arrhythmia requiring therapy, uncontrolled hypertension or congestive heart failure.
6. Arterial thrombotic or embolic events such as cerebrovascular accident (including ischemic attacks) or hemoptysis within 6 months before the first dose of study drug.
7. Venous thrombotic events (eg, deep vein thrombosis) or pulmonary arterial events (eg, pulmonary embolism) within 3 months before the first dose of study drug. Patients with venous thrombotic events ≥3 months before the first dose of study drug on stable anticoagulation therapy are eligible.
8. 12-lead electrocardiogram (ECG) demonstrating QT interval corrected by Fridericia's formula >450 ms in males or >470 ms in females at screening or history of long QT interval corrected syndrome.
9. Left ventricular ejection fraction (LVEF) <50% at screening.
10. Use of proton-pump inhibitors within 4 days prior to the first dose of study drug. Other medications that increase gastric pH, ie, histamine H2 receptor antagonists and antacids may be taken provided they are not administered within 2 hours before or after administration of study drug.
11. Use of strong or moderate inhibitors and inducers of cytochrome P450 (CYP) 3A4, including certain herbal medications (eg, St. John's Wort) and consumption of grapefruit or grapefruit juice within 14 days or 5 x the half-life (whichever is longer) prior to the first dose of study drug.
12. Use of known substrates or inhibitors of breast cancer resistance protein (BCRP) transporters within 14 days or 5 x the half-life (whichever is longer) prior to the first dose of study drug.
13. Major surgeries (eg, abdominal laparotomy) within 4 weeks of the first dose of study drug. Following major surgeries, >4 weeks prior to the first dose of study drug, all surgical wounds must be healed and free of infection or dehiscence.
14. Any other clinically significant comorbidities, such as uncontrolled pulmonary disease, active infection, or any other condition, which in the judgment of the Investigator, could compromise compliance with the protocol, interfere with interpretation of the study results, or predispose the patient to safety risks.
15. Known human immunodeficiency virus or hepatitis C infection only if the patient is taking medications that are excluded per protocol, active hepatitis B, or active hepatitis C infection.
16. If female, the patient is pregnant or lactating.
17. Known allergy or hypersensitivity to any component of the investigational drug product. Patients with a history of Stevens-Johnson syndrome on a prior TKI are excluded.
18. Gastrointestinal abnormalities including but not limited to:

    * inability to take oral medication
    * malabsorption syndromes
    * requirement for intravenous alimentation
19. Any active bleeding excluding hemorrhoidal or gum bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2022-05-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (15):
  - HonorHealth, Scottsdale, Arizona
  - University of Southern California - Norris, Los Angeles, California
  - UCLA, Los Angeles, California
  - Stanford, Stanford, California
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Georgia Cancer Specialists, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Columbia, New York, New York
  - MSKCC, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Alfred University, Melbourne, Australia
- University Hospital Leuven, Leuven, Belgium
- Canada (2):
  - Cross Cancer Center, Edmonton, Alberta
  - Princess Margaret Hospital, Toronto
- Helsinki University Central Hospital, Helsinki, Finland
- France (3):
  - Institut Bergonié, Bordeaux
  - Le Centre Léon Bérard, Lyon
  - Gustave-Roussy, Villejuif
- Germany (3):
  - Sarcoma Center Brandenburg, Brandenburg
  - University Hospital Essen, Essen
  - Universitätsmedizin Mannheim, Mannheim
- Italy (2):
  - Istituto Nazionale dei Tumori, Milan
  - Università Campus Bio-Medico di Roma, Rome
- Leiden University Medical Center, Leiden, Netherlands
- Maria Sklodowska-Curie Memorial Cancer Center, Warsaw, Poland
- NCC, Singapore, Singapore
- Spain (2):
  - Vall d'Hebron, Barcelona
  - Hospitalario Universitario Virgen del Rocío, Seville
- United Kingdom (2):
  - Royal Marsden, London
  - University of Sheffield, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schoffski P, George S, Heinrich MC, Zalcberg JR, Bauer S, Gelderblom H, Serrano C, Jones RL, Attia S, D'Amato G, Chi P, Reichardt P, Becker C, Shi K, Meade J, Ruiz-Soto R, Blay JY, von Mehren M. Patient-reported outcomes in individuals with advanced gastrointestinal stromal tumor treated with ripretinib in the fourth-line setting: analysis from the phase 3 INVICTUS trial. BMC Cancer. 2022 Dec 13;22(1):1302. doi: 10.1186/s12885-022-10379-9. PMID 36514034
- [Derived] Symcox M, Somaiah N. Ripretinib for advanced gastrointestinal stromal tumor: Plain language summary of the INVICTUS study. Future Oncol. 2021 Dec 1;17(36):5007-5012. doi: 10.2217/fon-2021-0803. Epub 2021 Oct 18. PMID 34661454
- [Derived] Blay JY, Serrano C, Heinrich MC, Zalcberg J, Bauer S, Gelderblom H, Schoffski P, Jones RL, Attia S, D'Amato G, Chi P, Reichardt P, Meade J, Shi K, Ruiz-Soto R, George S, von Mehren M. Ripretinib in patients with advanced gastrointestinal stromal tumours (INVICTUS): a double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Oncol. 2020 Jul;21(7):923-934. doi: 10.1016/S1470-2045(20)30168-6. Epub 2020 Jun 5. PMID 32511981
- See also: Deciphera Company Website — http://www.deciphera.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient enrolled on 27 Feb 2018, with the last patient in (LPI) on 16 Nov 2018. The study is ongoing; Data cutoff date of 31 May 2019. Of the 129 patients enrolled in the double-blind period (ITT population), 85 patients were randomized to the ripretinib arm and 44 patients were randomized to the placebo arm.
Groups:
- Ripretinib: Ripretinib (150 mg) once daily in 28-day cycles until disease progression by Independent Radiologic Review (IRR) in patients with advanced gastrointestinal stromal tumors (GIST) who have received treatment with prior therapies (therapies must include treatment with imatinib, sunitinib, and regorafenib). Ripretinib vs. Placebo 2:1 ratio
- Placebo: Placebo once daily in 28-day cycles until disease progression by Independent Radiologic Review (IRR) in patients with advanced gastrointestinal stromal tumors (GIST) who have received treatment with prior therapies (therapies must include treatment with imatinib, sunitinib, and regorafenib). Ripretinib vs. Placebo 2:1 ratio
Period: Overall Study
Arm/Group | Ripretinib | Placebo
Started | 85 | 44 (1 patient was randomized but not dosed)
Completed (Completed patients of the double-blind period are those that have entered the open-label period, or discontinued treatment due to death or confirmed progressive disease by IRR as of the cutoff of May 31, 2019.) | 46 | 35
Not Completed | 39 | 9

BASELINE CHARACTERISTICS:
Population: The baseline analysis population was the intent-to-treat (ITT) population, defined as those who signed the ICF and were randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Ripretinib | Placebo | Total
Number analyzed (Participants) | 85 | 44 | 129
Age, Customized [Count of Participants; unit: Participants]
  Age Category (years): 18 - 64 Years | 57 | 22 | 79
  Age Category (years): 65 - 74 Years | 20 | 12 | 32
  Age Category (years): 75 Years or Older | 8 | 10 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 18 | 56
  Male | 47 | 26 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 76 | 38 | 114
  Unknown or Not Reported | 8 | 6 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 4 | 5 | 9
  Race: Black or African American | 8 | 2 | 10
  Race: White | 64 | 33 | 97
  Race: Not Reported | 8 | 4 | 12
  Race: Other | 1 | 0 | 1
Region [Count of Participants; unit: Participants]
  US | 40 | 20 | 60
  Non-US | 45 | 24 | 69
Number of Prior Systemic Anticancer Treatments [Count of Participants; unit: Participants]
  3 | 54 | 27 | 81
  ≥ 4 | 31 | 17 | 48

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time interval between the date of randomization and the earliest documented evidence of the first disease progression based on the independent radiologic review or death due to any cause on initially assigned study treatment, whichever comes earlier, assessed at 26, 39, and 52 weeks.
Time Frame: From date of randomization to the earliest date of disease progression or death from any cause [through database cutoff 31-May-2019 (up to approximately 15 months)].
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Weeks
Groups:
- Ripretinib: Ripretinib (150 mg) once daily in 28-day cycles until disease progression by Independent Radiologic Review (IRR) in patients with advanced gastrointestinal stromal tumors (GIST) who have received treatment with prior therapies (therapies must include treatment with imatinib, sunitinib, and regorafenib).
- Placebo: Placebo once daily in 28-day cycles until disease progression by Independent Radiologic Review (IRR) in patients with advanced gastrointestinal stromal tumors (GIST) who have received treatment with prior therapies (therapies must include treatment with imatinib, sunitinib, and regorafenib).
Arm/Group | Ripretinib | Placebo
Number analyzed (Participants) | 85 | 44
Weeks | 27.6 [20.0 to 29.9] | 4.1 [4.0 to 7.3]
Statistical Analysis 1: Comparison: Ripretinib vs Placebo; Test type: Superiority; p < 0.0001, Log Rank — Two-sided P-value; Strata: prior lines of therapy (3 versus ≥4); ECOG (0 versus 1 or 2); Hazard Ratio, log = 0.15, 95% CI 2-sided [0.09 to 0.25] — Ripretinib: Placebo; based on stratified Cox Proportional Hazards Regression Model using randomization stratification factors [prior lines of therapy (3 versus ≥4); ECOG (0 versus 1 or 2)]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: The percentage of patients with a confirmed complete response or PR (CR: Disappearance of all target lesions and non-target lesions (if present at baseline); all lymph nodes must be non-pathological in size) or partial response (PR: >=30% decrease in the Sum of Diameters of target lesions and non-target lesions non-PD or NE or none at baseline; or target lesions CR and non-target lesions non-CR/Non-PD or NE) based on the independent radiologic review and during the initially assigned study treatment. To be assigned a status of a CR or PR, changes in tumor measurements must be confirmed by repeat CT or MRI assessments that must be performed at least 4 weeks after the criteria for response are first met.
Time Frame: as for outcome 1
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ripretinib | Placebo
Number analyzed (Participants) | 85 | 44
Percentage of Participants | 9.4 [4.2 to 17.7] | 0 [0.0 to 8.0]
Statistical Analysis 1: Comparison: Ripretinib vs Placebo; Test type: Superiority; p = 0.0504, Fisher Exact — Two-sided P-value

3. Secondary Outcome: Time to Tumor Progression (TTP) Based on Independent Radiologic Review
Description: TTP is defined as the interval between the date of randomization and the earliest documented evidence of disease progression based on the independent radiologic review.
Time Frame: From date of randomization to the earliest date of disease progression [through database cutoff 31-May-2019 (up to approximately 15 months)].
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ripretinib | Placebo
Number analyzed (Participants) | 85 | 44
Weeks | 28 [20.0 to 36.4] | 4.1 [4.0 to 7.6]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the interval between the date of randomization until the date of death or the date of last follow-up.
Time Frame: From the date of randomization to the date of death from any cause [through database cutoff 31-May-2019 (up to approximately 15 months)].
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Ripretinib | Placebo
Number analyzed (Participants) | 85 | 44
weeks | 65.6 [53.6 to 65.6] | 28.6 [17.9 to 50.4]
Statistical Analysis 1: Comparison: Ripretinib vs Placebo; Test type: Superiority; p = 0.0004, Log Rank — Not evaluated for statistical significance as a result of the sequential testing procedure for the secondary endpoints of ORR and OS; Strata: prior lines of therapy (3 versus ≥4); ECOG (0 versus 1 or 2); Hazard Ratio (HR) = 0.36, 95% CI 2-sided [0.21 to 0.62] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Quality of Life & Disease-Related Symptoms - European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire for Cancer 30-Item - Role Functioning
Description: Changes from baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire for Cancer 30-item - Role Functioning. For the ripretinib arm the minimum and maximum for the outcome were -67 to 67; the placebo arm had a range of -83 to 67. The higher value represents a higher quality of life in disease-related symptoms.
Time Frame: From the date of randomization (Baseline) to Cycle 2 Day 1 (Month 2)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ripretinib | Placebo
Number analyzed (Participants) | 85 | 43
units on a scale | 3.5 (27.31) | -17.1 (30.28)
Statistical Analysis 1: Comparison: Ripretinib vs Placebo; Test type: Superiority; p = 0.001, ANCOVA — Not evaluated for statistical significance as a result of the sequential testing procedure for the secondary endpoints of ORR, OS, and QOL; Factors: prior lines of therapy (3 versus ≥4); ECOG (0 versus 1 or 2)

6. Secondary Outcome: Quality of Life & Disease-Related Symptoms - Physical Functioning
Description: Changes from baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire for Cancer 30-Item - Physical Functioning. For the ripretinib arm, the minimum and maximum for the outcome were -33 to 53; the placebo arm had a range of -47 to 20. The higher value represents a higher quality of life in disease-related symptoms.
Time Frame: From the date of randomization (Baseline) to Cycle 2 Day 1 (Month 2)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ripretinib | Placebo
Number analyzed (Participants) | 85 | 43
units on a scale | 1.6 (16.03) | -8.9 (19.28)
Statistical Analysis 1: Comparison: Ripretinib vs Placebo; Test type: Superiority; p = 0.004, ANCOVA — [p-value comment as in outcome 5, analysis 1]; Factors: prior lines of therapy (3 versus ≥4); ECOG (0 versus 1 or 2)

7. Secondary Outcome: Quality of Life & Disease-Related Symptoms - EuroQol Visual Analogue Scale
Description: Change from baseline in EuroQol Visual Analogue Scale. For the ripretinib arm the minimum and maximum for the outcome were -43 to 91; the placebo arm had a range of -68 to 23. The higher value represents a higher quality of life in disease-related symptoms.
Time Frame: From the date of randomization (Baseline) to Cycle 2 Day 1 (Month 2)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Ripretinib | Placebo
Number analyzed (Participants) | 85 | 43
Units on a Scale | 3.7 (20.36) | -8.9 (19.31)
Statistical Analysis 1: Comparison: Ripretinib vs Placebo; Test type: Superiority; p = 0.004, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: After Administration of the first dose of study drug and through 30 days after the last dose of study drug. A median of 28 weeks per participant for the ripretinib arm, and a median of 10 weeks per participant for the placebo arm.
Description: Treatment-Emergent Adverse Events (TEAEs) are defined as any adverse event (all grades) that occurs after administration of the first dose of study drug and through 30 days after the last dose of study drug (Safety Population).The median treatment duration of the safety population for ripretinib arm was 23.86 weeks and placebo was 6 weeks during the double-blind period.
Arm/Group | Ripretinib | Placebo
All-Cause Mortality (participants affected / at risk) | 26/85 | 26/43
Serious Adverse Events (participants affected / at risk) | 26/85 | 19/43
Other Adverse Events (participants affected / at risk) | 84/85 | 42/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ripretinib (N=85) | Placebo (N=43)
Anemia (Blood and lymphatic system disorders) | 3 | 1
Abdominal Pain (Gastrointestinal disorders) | 4 | 2
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Death (General disorders) | 3 | 4
Cardiac Failure (Cardiac disorders) | 1 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 0
Fecaloma (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Fistula (Gastrointestinal disorders) | 1 | 1
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 1
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Perforation (Gastrointestinal disorders) | 0 | 1
General Physical Health Deterioration (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 1
Systemic Inflammatory Response Syndrome (General disorders) | 0 | 1
Liver Abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 1
Septic Shock (Infections and infestations) | 0 | 1
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood Bilirubin Increased (Investigations) | 1 | 0
Blood Creatinine Increased (Investigations) | 0 | 1
Hyperkaliemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatasemia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hallucinations, mixed (Psychiatric disorders) | 1 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 2
Urinary Retention (Renal and urinary disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Embolism (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ripretinib (N=85) | Placebo (N=43)
Anemia (Blood and lymphatic system disorders) | 12 | 8
Nausea (Gastrointestinal disorders) | 33 | 5
Abdominal Pain (Gastrointestinal disorders) | 31 | 13
Constipation (Gastrointestinal disorders) | 29 | 8
Diarrhea (Gastrointestinal disorders) | 24 | 6
Vomiting (Gastrointestinal disorders) | 18 | 3
Stomatitis (Gastrointestinal disorders) | 9 | 0
Abdominal Pain (Upper) (Gastrointestinal disorders) | 8 | 2
Dyspepsia (Gastrointestinal disorders) | 7 | 6
Fatigue (General disorders) | 36 | 10
Peripheral Edema (General disorders) | 14 | 3
Asthenia (General disorders) | 11 | 6
Pyrexia (General disorders) | 6 | 2
Weight Decreased (Investigations) | 16 | 5
Blood Bilirubin Increased (Investigations) | 14 | 0
Lipase Increased (Investigations) | 9 | 0
Aspartate Aminotransferase Increased (Investigations) | 6 | 2
Blood Alkaline Phosphatase Increased (Investigations) | 6 | 1
Alanine Aminotransferase Increased (Investigations) | 5 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 23 | 9
Hypophosphatemia (Metabolism and nutrition disorders) | 9 | 0
Hypokalemia (Metabolism and nutrition disorders) | 5 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 27 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 13 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 8 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 8 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Headache (Nervous system disorders) | 16 | 2
Dizziness (Nervous system disorders) | 7 | 3
Peripheral Sensory Neuropathy (Nervous system disorders) | 6 | 1
Insomnia (Psychiatric disorders) | 8 | 6
Anxiety (Psychiatric disorders) | 7 | 4
Depression (Psychiatric disorders) | 6 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 44 | 2
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 18 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 11 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 5 | 1
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 5 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 5 | 0
Pruritus Generalized (Skin and subcutaneous tissue disorders) | 5 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 5 | 0
Hypertension (Vascular disorders) | 12 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither Institution nor Investigator will submit for publication or public disclosure any publication or disclosure based on the results of the Study until after the first to occur of (a) publication of the Multi-Center Clinical Trial results; (b) notification by Sponsor that the Multi-Center Clinical Trial submission is no longer planned; or (c) the 12 month anniversary of the completion or early termination of the Multi-Center Clinical Trial.

DOCUMENTS (2):
  • Study Protocol (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT03353753/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/53/NCT03353753/SAP_001.pdf